CLINICAL TRIAL: NCT02961985
Title: Myokardinfarkt-Register Des Saarlandes (MIR-SL)
Brief Title: Myocardial Infarction Register of the Saarland
Acronym: MIR-SL
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Ministry of Social Affairs, Health, Women and Family of Saarland (Unknown)
Responsible Party: Sponsor
Other Study IDs: MIR-SL
Record Dates: First submitted 2016-09-05; First posted 2016-11-11 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Myocardial Infarction Register Saarland (MIR-SL), is intended to collect data about the treatment of patients suffering from ST-elevation myocardial infarction (STEMI). It aims to provide current data on the implementation of guidelines for both, the interventional and adjuvant drug therapy of STEMI in daily clinical practice in the Saarland.

DETAILED DESCRIPTION:
The Myocardial Infarction Register Saarland (MIR-SL), is intended to collect data about the treatment of patients suffering from ST-elevation myocardial infarction (STEMI). It aims to provide current data on the implementation of guidelines for both, the interventional and adjuvant drug therapy of STEMI in daily clinical practice in the Saarland.

In order to obtain representative data for the Saarland, preferably all consecutive patients should be documented comprehensively in the University Hospital of the Saarland, the non-university hospitals with cardiac catheterization laboratory as well as in hospitals without cardiac catheterization laboratory .

MIR-SL is attended by all 22 hospitals in Saarland, that treat patients with acute STEMI. A follow-up will be carried out after three months, 12 months and five years.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent

Exclusion Criteria:

* age < 18 years
* missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a hospital in the Saarland region with ST elevation myocardial infarction, in the last 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Rate of reperfusion therapies | 24 hours
  Describe hospital daily routine in Germany

SECONDARY OUTCOMES:
Time before reperfusion therapy | 24 hours
  pre-hospital time, intrahospital time, transfer time
In-hospital mortality | 24 hours
  Describe mortality before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Anselm K. Gitt, Dr., Principal Investigator — Stiftung Institut fuer Herzinfarktforschung
Locations (3):
- Germany (3):
  - Klinikum Saarbruecken, Saarbrücken, Saarland
  - Marienhaus Klinikum Saarlouis-Dillingen, Dillingen
  - Universitaetsklinikum des Saarlandes, Homburg

IPD SHARING:
Plan to Share IPD: No